CLINICAL TRIAL: NCT06957704
Title: Evaluation of the Efficacy and Safety of Subcutaneous Ketamine in the Treatment of Depressive Episode With Suicidal Ideation and/or Behavior in Adolescents
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Sheila Cavalcante Caetano, Professor; Post doctor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 82712924300005505
Record Dates: First submitted 2025-03-29; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-03

CONDITIONS: Depressive Disorder; Suicidal Ideas
Keywords: Adolescent; Ketamine; Major Depressive Disorder; Midazolam
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (Experimental): Participants were randomly by assigned. ketamine will be used as an adjunctive treatment at an initial dose of 0.5 mg/kg, administered subcutaneously twice weekly for four weeks under double-blind conditions. Dose adjustments between 0.5 to 1.0 mg/kg may occur based on patient response and tolerability.
  Interventions: Drug: ketamine
- Midazolam (Placebo Comparator): For the placebo group, midazolam will be administered subcutaneously at a dose of 1 mg diluted in 5 ml of 0.9% saline, twice weekly for four consecutive weeks, also under double-blind conditions.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: ketamine — Ketamine will be administered as adjunctive therapy at an initial dose of 0.5 mg/kg via subcutaneous injection, twice weekly for four weeks, under double-blind conditions. Dose adjustments between 0.5 and 1.0 mg/kg will be based on depressive symptoms, efficacy, and tolerability. All procedures will occur at the Ketamine Clinic of Federal University of São Paulo.
  Arms: Ketamine
Drug: Midazolam — Midazolam will be administered subcutaneously twice weekly for four consecutive weeks, also under double-blind conditions. The subject will be monitored continuously during the procedure, and every hour for three hours after the infusion.
  Arms: Midazolam

SUMMARY:
Evaluate the efficacy and safety of subcutaneous ketamine added to usual treatment in the management of depressive episodes with suicidal ideation or behavior in adolescent patients, compared to usual treatment added to placebo (midazolam).

DETAILED DESCRIPTION:
Depression affects approximately 8% of adolescents, with an estimated 60% showing inadequate response to current standard treatments. Ketamine, a glutamatergic modulator, has demonstrated efficacy in adults with treatment-resistant depression and has shown promising preliminary results in adolescent populations. This Phase III, randomized, double-blind, placebo-controlled clinical trial aims to evaluate the efficacy and safety of subcutaneous ketamine as an adjunctive treatment for adolescents experiencing a major depressive episode with active suicidal ideation and/or behavior.

Participants will be randomized into two parallel groups to receive either subcutaneous ketamine (0.5 to 1 mg/kg) or an active placebo (1 mg midazolam diluted in 5 ml of 0.9% saline), administered twice weekly for four weeks. All participants will continue their usual treatment regimens. A two-week post-treatment follow-up period will be conducted to assess the persistence of effects and monitor safety outcomes.

Clinical assessments include diagnostic and symptom severity scales validated for pediatric populations. The efficacy will be primarily measured by depression remission and response, while safety will be assessed via adverse event monitoring and clinical examination. The trial will include 30 participants per group, providing 80% power to detect a clinically significant difference of 8.7 points on the Montgomery-Åsberg Depression Rating Scale (MADRS) between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age between 12 and 19 years.
* Diagnosis of Major Depressive Episode, unipolar, made through the Schedule for Affective Disorders and Schizophrenia for School-Age Children (K-SADS-PL) administered by experienced evaluators, using DSM-5 criteria.
* Under usual treatment for Major Depressive Episode, including clinically indicated psychopharmacological treatment and/or psychosocial treatment at one of the two collaborating clinics (DICA and Conversas de Vida / Unifesp).
* Score ≥ 25 on the MADRS (Montgomery-Åsberg Depression Rating Scale).
* Score ≥ 28 on the CDRS (Children Depression Rating Scale).
* Score ≥ 2 on the Columbia Suicide Severity Rating Scale (C-SSRS).
* History of suicide attempt or significant suicidal ideation or planning with a plan or intention requiring emergency evaluation in the last 30 days.

Exclusion Criteria:

* Presence of the following psychiatric comorbidities: Autism Spectrum Disorder, Bipolar Disorder, Schizophrenia, Schizoaffective Disorder, or psychiatric disorder secondary to physical illness, and history of ketamine or other substance abuse or dependence in the last 6 months.
* Presence of Intellectual Disability (assessed by IQ testing).
* Presence of the following clinical comorbidities: history of myocardial infarction, congenital heart disease, decompensated cardiac arrhythmia, decompensated hypertension, porphyria, stroke, brain trauma with loss of consciousness, intracranial hypertension, hydrocephalus, central nervous system tumors, or central nervous system abnormalities.
* Previous treatment for depression with esketamine.
* Allergy to esketamine.
* If female: pregnancy or breastfeeding.

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Montgomery-Asberg Rating Scale (MADRS) Total Score at 24 Hours Post First Dose | Baseline (predose) and 24 hours post first dose
  The Montgomery-Åsberg Depression Rating Scale (MADRS) has a minimum score of 0 and a maximum score of 60; higher scores indicate worse depression. The primary efficacy endpoint of ketamine will be evaluated as follows:
  * Remission: Total score on the MADRS ≤ 12
  * Response: A reduction of more than 50% in the total MADRS score.
  * Lack of response: A reduction of less than 50% in the baseline MADRS scores.

SECONDARY OUTCOMES:
Remission and Response of Suicidal Ideation and Behavior Assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline (predose) and 24 hours post first dose
  The Columbia-Suicide Severity Rating Scale (C-SSRS) has a range from 0 to 5, where higher scores indicate greater severity of suicidal ideation or behavior.
  Secondary Efficacy Endpoint:
  * Remission of Suicide Risk: C-SSRS score = 0
  * Response: A 50% or greater improvement in the C-SSRS score.

REFERENCES:
- [Background] Zhou Y, Lan X, Wang C, Zhang F, Liu H, Fu L, Li W, Ye Y, Hu Z, Chao Z, Ning Y. Effect of Repeated Intravenous Esketamine on Adolescents With Major Depressive Disorder and Suicidal Ideation: A Randomized Active-Placebo-Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2024 May;63(5):507-518. doi: 10.1016/j.jaac.2023.05.031. Epub 2023 Jul 4. PMID 37414272
- [Background] Wilkinson ST, Ballard ED, Bloch MH, Mathew SJ, Murrough JW, Feder A, Sos P, Wang G, Zarate CA Jr, Sanacora G. The Effect of a Single Dose of Intravenous Ketamine on Suicidal Ideation: A Systematic Review and Individual Participant Data Meta-Analysis. Am J Psychiatry. 2018 Feb 1;175(2):150-158. doi: 10.1176/appi.ajp.2017.17040472. Epub 2017 Oct 3. PMID 28969441
- [Background] Willner P, Hale AS, Argyropoulos S. Dopaminergic mechanism of antidepressant action in depressed patients. J Affect Disord. 2005 May;86(1):37-45. doi: 10.1016/j.jad.2004.12.010. PMID 15820269
- [Background] Vecchia DD, Kanazawa LKS, Wendler E, de Almeida Soares Hocayen P, Bruginski E, Campos FR, Stern CAJ, Vital MABF, Miyoshi E, Wohr M, Schwarting RKW, Andreatini R. Effects of ketamine on vocal impairment, gait changes, and anhedonia induced by bilateral 6-OHDA infusion into the substantia nigra pars compacta in rats: Therapeutic implications for Parkinson's disease. Behav Brain Res. 2018 Apr 16;342:1-10. doi: 10.1016/j.bbr.2017.12.041. Epub 2018 Jan 4. PMID 29307665
- [Background] Vazquez, D. A., Caetano, S., Schlegel, R., Lourenço, E., Nemi, A., Slemian, A., & Sanchez, Z. M. (2021). Schoolless life and the mental health of public-school students during the Covid-19 pandemic. In SciELO Preprints. https://doi.org/10.1590/SciELOPreprints.2329
- [Background] Surjan J, Grossi JD, Del Porto JA, Delfino RS, de Oliveira Cerqueira R, Lucchese AC, Magalhaes E, Del Sant LC, Tuena MA, Nakahira C, Fava VAR, Steglich MS, Abdo GL, Barbosa MG, Sarin LM, Lacerda ALT. Efficacy and Safety of Subcutaneous Esketamine in the Treatment of Suicidality in Major Depressive Disorder and Bipolar Depression. Clin Drug Investig. 2022 Oct;42(10):865-873. doi: 10.1007/s40261-022-01193-z. Epub 2022 Aug 31. PMID 36044154
- [Background] Snaith RP, Hamilton M, Morley S, Humayan A, Hargreaves D, Trigwell P. A scale for the assessment of hedonic tone the Snaith-Hamilton Pleasure Scale. Br J Psychiatry. 1995 Jul;167(1):99-103. doi: 10.1192/bjp.167.1.99. PMID 7551619
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Scheuing L, Chiu CT, Liao HM, Chuang DM. Antidepressant mechanism of ketamine: perspective from preclinical studies. Front Neurosci. 2015 Jul 21;9:249. doi: 10.3389/fnins.2015.00249. eCollection 2015. PMID 26257598
- [Background] Saland SK, Schoepfer KJ, Kabbaj M. Hedonic sensitivity to low-dose ketamine is modulated by gonadal hormones in a sex-dependent manner. Sci Rep. 2016 Feb 18;6:21322. doi: 10.1038/srep21322. PMID 26888470
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Background] Robbins TW, Everitt BJ. Neurobehavioural mechanisms of reward and motivation. Curr Opin Neurobiol. 1996 Apr;6(2):228-36. doi: 10.1016/s0959-4388(96)80077-8. PMID 8725965
- [Background] Rhee TG, Shim SR, Forester BP, Nierenberg AA, McIntyre RS, Papakostas GI, Krystal JH, Sanacora G, Wilkinson ST. Efficacy and Safety of Ketamine vs Electroconvulsive Therapy Among Patients With Major Depressive Episode: A Systematic Review and Meta-analysis. JAMA Psychiatry. 2022 Dec 1;79(12):1162-1172. doi: 10.1001/jamapsychiatry.2022.3352. PMID 36260324
- [Background] Poznanski EO, Cook SC, Carroll BJ. A depression rating scale for children. Pediatrics. 1979 Oct;64(4):442-50. PMID 492809
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Parsaik AK, Singh B, Khosh-Chashm D, Mascarenhas SS. Efficacy of Ketamine in Bipolar Depression: Systematic Review and Meta-analysis. J Psychiatr Pract. 2015 Nov;21(6):427-35. doi: 10.1097/PRA.0000000000000106. PMID 26554325
- [Background] Nutt D, Demyttenaere K, Janka Z, Aarre T, Bourin M, Canonico PL, Carrasco JL, Stahl S. The other face of depression, reduced positive affect: the role of catecholamines in causation and cure. J Psychopharmacol. 2007 Jul;21(5):461-71. doi: 10.1177/0269881106069938. Epub 2006 Oct 18. PMID 17050654
- [Background] Murrough JW, Abdallah CG, Mathew SJ. Targeting glutamate signalling in depression: progress and prospects. Nat Rev Drug Discov. 2017 Jul;16(7):472-486. doi: 10.1038/nrd.2017.16. Epub 2017 Mar 17. PMID 28303025
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] March J, Karayal O, Chrisman A: CAPTN: The pediatric adverse event rating scale. Boston: Scientific Proceedings of the Annual Meeting of the American Academy of Child and Adolescent Psychiatry; 2007
- [Background] Maguire L, Bullard T, Papa L. Ketamine for acute suicidality in the emergency department: A systematic review. Am J Emerg Med. 2021 May;43:54-58. doi: 10.1016/j.ajem.2020.12.088. Epub 2021 Jan 14. PMID 33524683
- [Background] Lucchese AC, Sarin LM, Magalhaes EJM, Del Sant LC, B Puertas C, Tuena MA, Nakahira C, Fava VA, Delfino R, Surjan J, Steiglich MS, Barbosa M, Abdo G, Cohrs FM, Liberatori A, Del Porto JA, Lacerda AL, B Andreoli S. Repeated subcutaneous esketamine for treatment-resistant depression: Impact of the degree of treatment resistance and anxiety comorbidity. J Psychopharmacol. 2021 Feb;35(2):142-149. doi: 10.1177/0269881120978398. Epub 2021 Jan 9. PMID 33427015
- [Background] Loo CK, Galvez V, O'Keefe E, Mitchell PB, Hadzi-Pavlovic D, Leyden J, Harper S, Somogyi AA, Lai R, Weickert CS, Glue P. Placebo-controlled pilot trial testing dose titration and intravenous, intramuscular and subcutaneous routes for ketamine in depression. Acta Psychiatr Scand. 2016 Jul;134(1):48-56. doi: 10.1111/acps.12572. Epub 2016 Mar 30. PMID 27028832
- [Background] Li N, Liu RJ, Dwyer JM, Banasr M, Lee B, Son H, Li XY, Aghajanian G, Duman RS. Glutamate N-methyl-D-aspartate receptor antagonists rapidly reverse behavioral and synaptic deficits caused by chronic stress exposure. Biol Psychiatry. 2011 Apr 15;69(8):754-61. doi: 10.1016/j.biopsych.2010.12.015. Epub 2011 Feb 3. PMID 21292242
- [Background] Lally N, Nugent AC, Luckenbaugh DA, Niciu MJ, Roiser JP, Zarate CA Jr. Neural correlates of change in major depressive disorder anhedonia following open-label ketamine. J Psychopharmacol. 2015 May;29(5):596-607. doi: 10.1177/0269881114568041. Epub 2015 Feb 17. PMID 25691504
- [Background] Lally N, Nugent AC, Luckenbaugh DA, Ameli R, Roiser JP, Zarate CA. Anti-anhedonic effect of ketamine and its neural correlates in treatment-resistant bipolar depression. Transl Psychiatry. 2014 Oct 14;4(10):e469. doi: 10.1038/tp.2014.105. PMID 25313512
- [Background] Kokkinou M, Ashok AH, Howes OD. The effects of ketamine on dopaminergic function: meta-analysis and review of the implications for neuropsychiatric disorders. Mol Psychiatry. 2018 Jan;23(1):59-69. doi: 10.1038/mp.2017.190. Epub 2017 Oct 3. PMID 28972576
- [Background] Kim S, Rush BS, Rice TR. A systematic review of therapeutic ketamine use in children and adolescents with treatment-resistant mood disorders. Eur Child Adolesc Psychiatry. 2021 Oct;30(10):1485-1501. doi: 10.1007/s00787-020-01542-3. Epub 2020 May 8. PMID 32385697
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Koretz D, Merikangas KR, Rush AJ, Walters EE, Wang PS; National Comorbidity Survey Replication. The epidemiology of major depressive disorder: results from the National Comorbidity Survey Replication (NCS-R). JAMA. 2003 Jun 18;289(23):3095-105. doi: 10.1001/jama.289.23.3095. PMID 12813115
- [Background] Kaufman J, Birmaher B, Brent D, Rao U, Flynn C, Moreci P, Williamson D, Ryan N. Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL): initial reliability and validity data. J Am Acad Child Adolesc Psychiatry. 1997 Jul;36(7):980-8. doi: 10.1097/00004583-199707000-00021. PMID 9204677
- [Background] Jaen-Varas D, Mari JJ, Asevedo E, Borschmann R, Diniz E, Ziebold C, Gadelha A. The association between adolescent suicide rates and socioeconomic indicators in Brazil: a 10-year retrospective ecological study. Braz J Psychiatry. 2019 Feb 18;41(5):389-395. doi: 10.1590/1516-4446-2018-0223. eCollection 2019. PMID 30785539
- [Background] Greenberg PE, Fournier AA, Sisitsky T, Pike CT, Kessler RC. The economic burden of adults with major depressive disorder in the United States (2005 and 2010). J Clin Psychiatry. 2015 Feb;76(2):155-62. doi: 10.4088/JCP.14m09298. PMID 25742202
- [Background] Glue P, Medlicott NJ, Harland S, Neehoff S, Anderson-Fahey B, Le Nedelec M, Gray A, McNaughton N. Ketamine's dose-related effects on anxiety symptoms in patients with treatment refractory anxiety disorders. J Psychopharmacol. 2017 Oct;31(10):1302-1305. doi: 10.1177/0269881117705089. Epub 2017 Apr 26. PMID 28441895
- [Background] George D, Galvez V, Martin D, Kumar D, Leyden J, Hadzi-Pavlovic D, Harper S, Brodaty H, Glue P, Taylor R, Mitchell PB, Loo CK. Pilot Randomized Controlled Trial of Titrated Subcutaneous Ketamine in Older Patients with Treatment-Resistant Depression. Am J Geriatr Psychiatry. 2017 Nov;25(11):1199-1209. doi: 10.1016/j.jagp.2017.06.007. Epub 2017 Jun 13. PMID 28739263
- [Background] Garcia LS, Comim CM, Valvassori SS, Reus GZ, Barbosa LM, Andreazza AC, Stertz L, Fries GR, Gavioli EC, Kapczinski F, Quevedo J. Acute administration of ketamine induces antidepressant-like effects in the forced swimming test and increases BDNF levels in the rat hippocampus. Prog Neuropsychopharmacol Biol Psychiatry. 2008 Jan 1;32(1):140-4. doi: 10.1016/j.pnpbp.2007.07.027. Epub 2007 Aug 8. PMID 17884272
- [Background] Garcia LS, Comim CM, Valvassori SS, Reus GZ, Stertz L, Kapczinski F, Gavioli EC, Quevedo J. Ketamine treatment reverses behavioral and physiological alterations induced by chronic mild stress in rats. Prog Neuropsychopharmacol Biol Psychiatry. 2009 Apr 30;33(3):450-5. doi: 10.1016/j.pnpbp.2009.01.004. Epub 2009 Jan 21. PMID 19439250
- [Background] Galvez V, O'Keefe E, Cotiga L, Leyden J, Harper S, Glue P, Mitchell PB, Somogyi AA, DeLory A, Loo CK. Long-lasting effects of a single subcutaneous dose of ketamine for treating melancholic depression: a case report. Biol Psychiatry. 2014 Aug 1;76(3):e1-2. doi: 10.1016/j.biopsych.2013.12.010. Epub 2014 Jan 3. No abstract available. PMID 24507509
- [Background] Friedrich MJ. Depression Is the Leading Cause of Disability Around the World. JAMA. 2017 Apr 18;317(15):1517. doi: 10.1001/jama.2017.3826. No abstract available. PMID 28418490
- [Background] Fava VAR, Sarin LM, Lucchese AC, Del Sant L, Magalhaes E, Delfino RS, Tuena MA, Nakahira C, Jackowski AP, Abdo G, Surjan J, Steiglich M, Barbosa MG, Porto JAD, Lacerda ALT, Cogo-Moreira H. The probability of response after each subcutaneous injection of esketamine in treatment-resistant depression. Rev Psiquiatr Salud Ment (Engl Ed). 2020 Oct 16:S1888-9891(20)30117-8. doi: 10.1016/j.rpsm.2020.10.003. Online ahead of print. English, Spanish. PMID 33075541
- [Background] Dwyer JB, Landeros-Weisenberger A, Johnson JA, Londono Tobon A, Flores JM, Nasir M, Couloures K, Sanacora G, Bloch MH. Efficacy of Intravenous Ketamine in Adolescent Treatment-Resistant Depression: A Randomized Midazolam-Controlled Trial. Am J Psychiatry. 2021 Apr 1;178(4):352-362. doi: 10.1176/appi.ajp.2020.20010018. Epub 2021 Mar 3. PMID 33653121
- [Background] Duman RS, Aghajanian GK. Synaptic dysfunction in depression: potential therapeutic targets. Science. 2012 Oct 5;338(6103):68-72. doi: 10.1126/science.1222939. PMID 23042884
- [Background] Del Sant LC, Sarin LM, Magalhaes EJM, Lucchese AC, Tuena MA, Nakahira C, Fava VAR, Delfino R, Surjan J, Steiglich MS, Barbosa M, Abdo G, Cohrs FM, Liberatori A, Del Porto JA, Lacerda ALT, de Jesus Mari J. Effects of subcutaneous esketamine on blood pressure and heart rate in treatment-resistant depression. J Psychopharmacol. 2020 Oct;34(10):1155-1162. doi: 10.1177/0269881120922955. Epub 2020 Jul 8. PMID 32638662
- [Background] Delfino RS, Del-Porto JA, Surjan J, Magalhaes E, Sant LCD, Lucchese AC, Tuena MA, Nakahira C, Fava VAR, Steglich MS, Barbosa MG, Sarin LM, Lacerda ALT. Comparative effectiveness of esketamine in the treatment of anhedonia in bipolar and unipolar depression. J Affect Disord. 2021 Jan 1;278:515-518. doi: 10.1016/j.jad.2020.09.056. Epub 2020 Sep 15. PMID 33017679
- [Background] Cullen KR, Amatya P, Roback MG, Albott CS, Westlund Schreiner M, Ren Y, Eberly LE, Carstedt P, Samikoglu A, Gunlicks-Stoessel M, Reigstad K, Horek N, Tye S, Lim KO, Klimes-Dougan B. Intravenous Ketamine for Adolescents with Treatment-Resistant Depression: An Open-Label Study. J Child Adolesc Psychopharmacol. 2018 Sep;28(7):437-444. doi: 10.1089/cap.2018.0030. Epub 2018 Jul 13. PMID 30004254
- [Background] Caye A, Kieling RR, Rocha TB, Graeff-Martins AS, Geyer C, Krieger F, Manfro GG, Brentani H, Isolan L, Rosario MC, Grassi-Oliveira R, Caetano SC, Moriyama T, Rohde LA, Kieling C. Schedule for Affective Disorders and Schizophrenia for School-Age Children - Present and Lifetime Version (K-SADS-PL), DSM-5 update: translation into Brazilian Portuguese. Braz J Psychiatry. 2017 Oct-Dec;39(4):384-386. doi: 10.1590/1516-4446-2017-2317. No abstract available. PMID 29160533
- [Background] Cavenaghi VB, da Costa LP, Lacerda ALT, Hirata ES, Miguel EC, Fraguas R. Subcutaneous Ketamine in Depression: A Systematic Review. Front Psychiatry. 2021 May 28;12:513068. doi: 10.3389/fpsyt.2021.513068. eCollection 2021. PMID 34122156
- [Background] Boletim Epidemiológico número 33 da Coordenação-Geral de Doenças e Agravos Não Transmissíveis do Departamento de Análise em Saúde e Vigilância das Doenças Não Transmissíveis da Secretaria de Vigilância em Saúde (CGDANT/DASNT/SVS/MS): Oliveira RV. Coordenação-Geral de Saúde Mental Álcool e outras Drogas do Departamento de Ações Programáticas Estratégicas da Secretaria de Atenção Primária à Saúde (CGMAD/ DAPES/SAPS/MS): Ribeiro RB, Santos AF, Almeida L, Juliani LW. Coordenação de Saúde do Homem do Departamento de Ações Programáticas Estratégicas (COSAH/DAPES/SAPS/MS): Albuquerque FP. Universidade Federal de São Paulo (Unifesp): Caetano SC.
- [Background] Bodden DHM, Stikkelbroek Y, Dirksen CD. Societal burden of adolescent depression, an overview and cost-of-illness study. J Affect Disord. 2018 Dec 1;241:256-262. doi: 10.1016/j.jad.2018.06.015. Epub 2018 Jul 18. PMID 30138810
- [Background] Beck AT, Steer RA, Ranieri WF. Scale for Suicide Ideation: psychometric properties of a self-report version. J Clin Psychol. 1988 Jul;44(4):499-505. doi: 10.1002/1097-4679(198807)44:43.0.co;2-6. PMID 3170753
- [Background] Ballard ED, Wills K, Lally N, Richards EM, Luckenbaugh DA, Walls T, Ameli R, Niciu MJ, Brutsche NE, Park L, Zarate CA Jr. Anhedonia as a clinical correlate of suicidal thoughts in clinical ketamine trials. J Affect Disord. 2017 Aug 15;218:195-200. doi: 10.1016/j.jad.2017.04.057. Epub 2017 Apr 25. PMID 28477497
- [Background] Argyropoulos SV, Nutt DJ. Anhedonia revisited: is there a role for dopamine-targeting drugs for depression? J Psychopharmacol. 2013 Oct;27(10):869-77. doi: 10.1177/0269881113494104. Epub 2013 Jul 31. PMID 23904408
- [Background] Andrews G, Issakidis C, Sanderson K, Corry J, Lapsley H. Utilising survey data to inform public policy: comparison of the cost-effectiveness of treatment of ten mental disorders. Br J Psychiatry. 2004 Jun;184:526-33. doi: 10.1192/bjp.184.6.526. PMID 15172947
- [Background] Andrade C. Ketamine for Depression, 4: In What Dose, at What Rate, by What Route, for How Long, and at What Frequency? J Clin Psychiatry. 2017 Jul;78(7):e852-e857. doi: 10.4088/JCP.17f11738. PMID 28749092
- [Background] Alnefeesi Y, Chen-Li D, Krane E, Jawad MY, Rodrigues NB, Ceban F, Di Vincenzo JD, Meshkat S, Ho RCM, Gill H, Teopiz KM, Cao B, Lee Y, McIntyre RS, Rosenblat JD. Real-world effectiveness of ketamine in treatment-resistant depression: A systematic review & meta-analysis. J Psychiatr Res. 2022 Jul;151:693-709. doi: 10.1016/j.jpsychires.2022.04.037. Epub 2022 May 25. PMID 35688035
- [Background] Abdallah CG, Jackowski A, Salas R, Gupta S, Sato JR, Mao X, Coplan JD, Shungu DC, Mathew SJ. The Nucleus Accumbens and Ketamine Treatment in Major Depressive Disorder. Neuropsychopharmacology. 2017 Jul;42(8):1739-1746. doi: 10.1038/npp.2017.49. Epub 2017 Mar 8. PMID 28272497
- [Background] Abbar M, Demattei C, El-Hage W, Llorca PM, Samalin L, Demaricourt P, Gaillard R, Courtet P, Vaiva G, Gorwood P, Fabbro P, Jollant F. Ketamine for the acute treatment of severe suicidal ideation: double blind, randomised placebo controlled trial. BMJ. 2022 Feb 2;376:e067194. doi: 10.1136/bmj-2021-067194. PMID 35110300